CLINICAL TRIAL: NCT03381287
Title: A Randomized, Double Blind, Placebo Controlled, Multicenter, Multiple Ascending Dose Study to Evaluate the Safety and Tolerability of HTD1801 in Adults With Hypercholesterolemia
Brief Title: A Multiple Ascending Dose Study of HTD1801 in Adults With Hypercholesterolemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: HighTide Biopharma Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HTD1801.PCT004
Record Dates: First submitted 2017-12-18; First posted 2017-12-21 (Actual); Results first posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2022-08

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HTD1801 250 mg BID (Experimental): Subjects received 500 mg/day HTD1801
  Interventions: Drug: HTD1801 Tablets, 500 mg
- HTD1801 500 mg BID (Experimental): Subjects received 1000 mg/day HTD1801
  Interventions: Drug: HTD1801 Tablets, 1000 mg
- HTD1801 1000 mg BID (Experimental): Subjects received 2000 mg/day HTD1801
  Interventions: Drug: HTD1801 Tablets, 2000 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo to match 500 mg HTD1801; Drug: Placebo to match 1000 mg HTD1801; Drug: Placebo to match 2000 mg HTD1801

INTERVENTIONS:
Drug: HTD1801 Tablets, 500 mg — 500 mg/day (250 mg BID)
  Arms: HTD1801 250 mg BID
Drug: HTD1801 Tablets, 1000 mg — 1000 mg/day (500 mg BID)
  Arms: HTD1801 500 mg BID
Drug: HTD1801 Tablets, 2000 mg — 2000 mg/day (1000 mg BID)
  Arms: HTD1801 1000 mg BID
Drug: Placebo to match 500 mg HTD1801 — 2 tablets/day (1 tablet BID)
  Arms: Placebo
Drug: Placebo to match 1000 mg HTD1801 — 4 tablets/day (2 tablet BID)
  Arms: Placebo
Drug: Placebo to match 2000 mg HTD1801 — 8 tablets/day (4 tablet BID)
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multicenter, multiple ascending dose (MAD) study to evaluate the safety and tolerability, pharmacokinetic (PK), and pharmacodynamic (PD) profiles of HTD1801 in overweight to obese adults with hypercholesterolemia. There were 3 cohorts of dose levels as 500, 1000 and 2000 mg/day, with 16 subjects planned for each cohort randomized 3:1 to receive either HTD1801 or Placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent
2. Males or females aged 18 to 70 years old at the time of first dosing
3. Have a body mass index (BMI) of >25.0 and ≤ 45.0 kg/m2 at Screening
4. Have a documented history of hypercholesterolemia, defined as LDL-C ≥ 2.59 mmol/L

Exclusion Criteria:

1. The use of any anti-dyslipidemia agent within 28 days prior to dosing
2. History of a total cholesterol ≥ 10.35 mmol/L or triglyceride ≥ 11.3 mmol/L
3. History of a clinically significant cardiac arrhythmia or clinically significant abnormal ECG results at Screening
4. Significant peripheral or coronary vascular disease
5. Clinically significant abnormal blood pressure at Screening or Baseline, defined as supine blood pressure ≥160/100 mmHg, or ≤ 90/60 mmHg
6. Primary hypothyroidism (thyroid stimulating hormone [TSH] > upper limit or normal [ULN] and free T4 < lower limit of normal [LLN]), primary subclinical hypothyroidism (screening TSH > ULN and free T4 within normal limits [WNL]), or secondary hypothyroidism (screening TSH < LLN and free T4< LLN) at Screening
7. Glucose-6-phosphate dehydrogenase (G6PD) deficiency

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-04-13 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Di Bisceglie, MD,FACP,FAASLD, Study Director — HighTide Therapeutics USA, LLC
Locations (3):
- Australia (3):
  - Q-Pharm Pty Ltd., Herston, Queensland
  - CMAX Clinical Research Pty Ltd, Adelaide, South Australia
  - Linear Clinical Research, Nedlands, Western Australia

REFERENCES:
- [Derived] Di Bisceglie AM, Watts GF, Lavin P, Yu M, Bai R, Liu L. Pharmacokinetics and pharmacodynamics of HTD1801 (berberine ursodeoxycholate, BUDCA) in patients with hyperlipidemia. Lipids Health Dis. 2020 Nov 12;19(1):239. doi: 10.1186/s12944-020-01406-4. PMID 33183320

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | HTD1801 250 mg BID | HTD1801 500 mg BID | HTD1801 1000 mg BID
Started | 12 | 12 | 12 | 14
Completed | 12 | 11 | 12 | 12
Not Completed | 0 | 1 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- HTD1801 500 mg BID: Subjects received 1000 mg/day HTD1801
  HTD1801 Tablets, 1000mg: 1000 mg/day (500 mg BID)
- Total: Total of all reporting groups
Arm/Group | Placebo | HTD1801 250 mg BID | HTD1801 500 mg BID | HTD1801 1000 mg BID | Total
Number analyzed (Participants) | 12 | 12 | 12 | 14 | 50
Age, Continuous [Mean (Full Range); unit: years] | 53.4 [26 to 63] | 48.4 [27 to 70] | 54.3 [42 to 63] | 52.0 [22 to 70] | 52.0 [22 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 5 | 10 | 30
  Male | 3 | 6 | 7 | 4 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 12 | 12 | 14 | 50
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 11 | 11 | 12 | 13 | 47
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Treatment-Emergent Adverse Events (TEAEs)
Description: TEAEs are defined as any AEs that commenced on or after exposure to study drug or any pre-existing AE that worsened in either intensity or frequency after exposure to study drug.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | HTD1801 250 mg BID | HTD1801 500 mg BID | HTD1801 1000 mg BID
Number analyzed (Participants) | 12 | 12 | 12 | 14
Participants
  TEAE | 8 | 10 | 8 | 11
  Serious TEAE | 0 | 0 | 0 | 1
  Severe TEAE | 1 | 0 | 0 | 0
  Drug-related TEAEs | 4 | 2 | 7 | 6
  TEAEs leading to treatment interrupted or discontinued | 0 | 0 | 0 | 1

2. Secondary Outcome: Maximum Plasma Concentration (Cmax) of HTD1801 Components After Single-dose Oral Administration
Time Frame: 0. 0.25, 0.5, 1, 2, 3, 4, 8, 12 and 24 hours on Day 1
Population: Specific PK samples were excluded from the PK analysis dataset as they were identified to have outside the established stability range for frozen sample storage.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- HTD1801 250 mg: Subjects received a single 250 mg HTD1801 tablet administered orally
- HTD1801 500 mg: Subjects received two 250 mg HTD1801 tablet administered orally
- HTD1801 1000 mg: Subjects received four 250 mg HTD1801 tablet administered orally
Arm/Group | HTD1801 250 mg | HTD1801 500 mg | HTD1801 1000 mg
Number analyzed (Participants) | 12 | 12 | 14
ng/mL
  Berberine (BBR) | 0.390 (0.163) | 0.441 (0.286) | 0.865 (0.451)
  Ursodeoxycholic Acid (UDCA): number analyzed (Participants) | 12 | 10 | 14
  Ursodeoxycholic Acid (UDCA) | 923 (453) | 1900 (847) | 2900 (1520)

3. Secondary Outcome: Maximum Plasma Concentration (Cmax) of HTD1801 Components After Multiple-dose Oral Administration
Time Frame: 0. 0.25, 0.5, 1, 2, 3, 4, 8, 12 and 24 hours on Day 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- HTD1801 250 mg BID: Subjects received a single 250 mg HTD1801 tablet administered orally BID
- HTD1801 500 mg BID: Subjects received two 250 mg HTD1801 tablet administered orally BID
- HTD1801 1000 mg BID: Subjects received four 250 mg HTD1801 tablet administered orally BID
Arm/Group | HTD1801 250 mg BID | HTD1801 500 mg BID | HTD1801 1000 mg BID
Number analyzed (Participants) | 11 | 12 | 12
ng/mL
  Berberine (BBR) | 0.676 (0.231) | 1.510 (1.200) | 1.770 (1.310)
  Ursodeoxycholic Acid (UDCA): number analyzed (Participants) | 10 | 11 | 12
  Ursodeoxycholic Acid (UDCA) | 962 (275) | 1900 (825) | 3370 (966)

4. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of HTD1801 Components After Single-dose Oral Administration
Time Frame: 0. 0.25, 0.5, 1, 2, 3, 4, 8, 12 and 24 hours on Day 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | HTD1801 250 mg | HTD1801 500 mg | HTD1801 1000 mg
Number analyzed (Participants) | 12 | 12 | 14
hours
  Berberine (BBR) | 3.5 [2.0 to 8.25] | 4.0 [2.0 to 8.0] | 4.0 [3.0 to 12.0]
  Ursodeoxycholic Acid (UDCA): number analyzed (Participants) | 12 | 10 | 14
  Ursodeoxycholic Acid (UDCA) | 2.0 [0.50 to 4.0] | 3.0 [1.0 to 4.07] | 4.0 [1.0 to 8.0]

5. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of HTD1801 Components After Multiple-dose Oral Administration
Time Frame: 0. 0.25, 0.5, 1, 2, 3, 4, 8, 12 and 24 hours on Day 28
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | HTD1801 250 mg BID | HTD1801 500 mg BID | HTD1801 1000 mg BID
Number analyzed (Participants) | 11 | 12 | 12
hours
  Berberine (BBR) | 4.0 [0.0 to 4.0] | 4.0 [0.25 to 12.0] | 4.0 [2.0 to 12.0]
  Ursodeoxycholic Acid (UDCA): number analyzed (Participants) | 11 | 11 | 12
  Ursodeoxycholic Acid (UDCA) | 3.0 [2.0 to 12.0] | 4.0 [2.0 to 8.0] | 3.0 [0.0 to 4.03]

6. Secondary Outcome: Plasma Half-life of HTD1801 Components (T1/2) After Single-dose Oral Administration
Time Frame: 0.25, 0.5, 1, 2, 3, 4, 8, 12 and 24 hours on Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | HTD1801 250 mg | HTD1801 500 mg | HTD1801 1000 mg
Number analyzed (Participants) | 5 | 3 | 3
hours
  Berberine (BBR): number analyzed (Participants) | 5 | 2 | 3
  Berberine (BBR) | 9.04 (1.50) | 10.60 (2.51) | 7.79 (0.60)
  Ursodeoxycholic Acid (UDCA) | 2.79 (0.92) | 8.43 (11.30) | 5.24 (1.64)

7. Secondary Outcome: Plasma Half-life of HTD1801 Components (T1/2) After Multiple-dose Oral Administration
Time Frame: 0. 0.25, 0.5, 1, 2, 3, 4, 8, 12 and 24 hours on Day 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | HTD1801 250 mg BID | HTD1801 500 mg BID | HTD1801 1000 mg BID
Number analyzed (Participants) | 0 | 3 | 4
hours
  Berberine (BBR): number analyzed (Participants) | 0 | 0 | 0
  Ursodeoxycholic Acid (UDCA) |  | 7.60 (2.90) | 7.53 (2.78)

8. Secondary Outcome: Percent Change in Low-density Lipoprotein-Cholesterol (LDL-C) From Baseline to Day 28 Within and Between Treatment Groups
Time Frame: Baseline, Day 14, Day 28
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Placebo | HTD1801 250 mg BID | HTD1801 500 mg BID | HTD1801 1000 mg BID
Number analyzed (Participants) | 11 | 11 | 11 | 12
percentage change from baseline
  Percent Change from Baseline to Day 14 | 3.624 (11.9910) | -3.390 (8.3100) | -1.1550 (26.2682) | -9.296 (14.9090)
  Percent Change from Baseline to Day 28 | -3.585 (21.7628) | -7.674 (13.1407) | 0.372 (15.3368) | -9.767 (12.6763)

9. Secondary Outcome: Percent Change in Triglycerides From Baseline to Day 28 Within and Between Treatment Groups
Time Frame: Baseline, Day 14, Day 28
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Placebo | HTD1801 250 mg BID | HTD1801 500 mg BID | HTD1801 1000 mg BID
Number analyzed (Participants) | 12 | 12 | 12 | 14
percentage change from baseline
  Percent Change from Baseline to Day 14 | 1.724 (19.4047) | -5.788 (25.4470) | 12.798 (34.8867) | -2.240 (28.2301)
  Percent Change from Baseline to Day 28 | 36.778 (30.1113) | 7.684 (27.8053) | 25.882 (34.6145) | 6.256 (18.4114)

10. Secondary Outcome: Percent Change in Free-fatty Acids (FFA) From Baseline to Day 28 Within and Between Treatment Groups
Time Frame: Baseline, Day 14, Day 28
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Placebo | HTD1801 250 mg BID | HTD1801 500 mg BID | HTD1801 1000 mg BID
Number analyzed (Participants) | 9 | 5 | 12 | 10
percentage change from baseline
  Percent Change from Baseline to Day 14 | -41.743 (29.7652) | -38.672 (37.1275) | -41.295 (20.1601) | -32.192 (28.0350)
  Percent Change from Baseline to Day 28 | -33.153 (33.9741) | -46.458 (36.1597) | 47.246 (18.0392) | -34.382 (24.8417)

11. Secondary Outcome: Percent Change in Lipoprotein-A From Baseline to Day 28 Within and Between Treatment Groups
Time Frame: Baseline, Day 14, Day 28
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Placebo | HTD1801 250 mg BID | HTD1801 500 mg BID | HTD1801 1000 mg BID
Number analyzed (Participants) | 10 | 11 | 8 | 12
percentage change from baseline
  Percent Change from Baseline to Day 14 | -4.975 (27.7800) | -19.527 (22.0535) | 222.4113 (214.9631) | -13.034 (27.9322)
  Percent Change from Baseline to Day 28 | 10.582 (20.4217) | -11.239 (33.9248) | 242.570 (477.1207) | -21.916 (26.2907)

ADVERSE EVENTS:
Time Frame: 4 weeks
Groups:
- HTD1801 250 mg BID: Subjects received 500 mg/day HTD1801
  HTD1801 Tablets, 500mg: 500 mg/day (250 mg bid)
- HTD1801 1000 mg BID: Subjects received 2000 mg/day HTD1801
  HTD1801 Tablets, 2000mg: 2000 mg/day (1000 mg bid)
Arm/Group | Placebo | HTD1801 250 mg BID | HTD1801 500 mg BID | HTD1801 1000 mg BID
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 1/14
Other Adverse Events (participants affected / at risk) | 8/12 | 10/12 | 8/12 | 11/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=12) | HTD1801 250 mg BID (N=12) | HTD1801 500 mg BID (N=12) | HTD1801 1000 mg BID (N=14)
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatitis. (Hepatobiliary disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=12) | HTD1801 250 mg BID (N=12) | HTD1801 500 mg BID (N=12) | HTD1801 1000 mg BID (N=14)
Headache (Nervous system disorders) | 5 | 5 | 4 | 3
Dizziness (Nervous system disorders) | 0 | 2 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 1 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 2 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Change of bowel habit (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Viral pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0
Catheter site erythema (General disorders) | 0 | 0 | 0 | 1
Catheter site pain (General disorders) | 1 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 1 | 0 | 0
Ulcer (General disorders) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 3 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Tendon pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 1 | 0
Vascular pain (Vascular disorders) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-01-19): https://cdn.clinicaltrials.gov/large-docs/87/NCT03381287/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-09): https://cdn.clinicaltrials.gov/large-docs/87/NCT03381287/SAP_001.pdf